CLINICAL TRIAL: NCT04089449
Title: A Phase 1, Open-Label, Multicenter, Dose Escalation and Expansion Study of PRT811 in Subjects With Advanced Solid Tumors, CNS Lymphoma, and Recurrent High-Grade Gliomas
Brief Title: A Study of PRT811 in Participants With Advanced Solid Tumors, CNS Lymphoma and Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prelude Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRT811-01
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Advanced Solid Tumor; Recurrent Glioma
Keywords: PRMT5; PRMT5 Inhibitor
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PRT811 (Experimental): PRT811 will be administered orally
  Interventions: Drug: PRT811

INTERVENTIONS:
Drug: PRT811 — PRT811 will be administered orally

SUMMARY:
This is a Phase 1 dose-escalation study of PRT811, a protein arginine N-methyltransferase (PRMT) 5 inhibitor, in subjects with advanced cancers and high-grade gliomas who have exhausted available treatment options. The purpose of this study is to define a safe dose and schedule to be used in subsequent development of PRT811.

DETAILED DESCRIPTION:
This is a multicenter, open-label, dose-escalation, dose-expansion Phase 1 study of PRT811, a PRMT5 inhibitor, in subjects with advanced cancers without any approved or available treatment options including solid tumors, CNS lymphoma, and /or high-grade gliomas. The study will consist of 2 parts, a dose escalation part evaluating subjects with advanced solid tumors, CNS lymphoma, and/or high-grade glioma and a cohort expansion part which will evaluate the safety and efficacy of PRT811 in subjects with advanced solid tumors, and glioblastoma multiforme. For subjects, the study will include a screening phase, a treatment phase, and a post treatment follow-up phase. An end-of-study visit will be conducted within 30 days after the last dose of PRT811.

ELIGIBILITY:
Inclusion Criteria:

* Malignancies that are refractory to or intolerant of established therapies known to provide clinical benefit for the malignancy in question, or in the opinion of the Investigator, not be a candidate for such therapies
* Subjects must have recovered from the effects of any prior investigational system therapies
* For subjects with recurrent high-grade glioma or GBM, must have biopsy proven evidence (WHO Grade III or IV) and received external bean fractionated radiotherapy and at least 2 cycles of adjuvant temozolomide chemotherapy. Mutant Glioma must comply with biomarker defined enrollment criterias.
* For biomarker-selected solid tumors: must meet enrollment criteria
* Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1
* Adequate organ function (bone marrow, hepatic, renal, cardiovascular)
* Female subjects of childbearing potential must have a negative pregnancy test within 7 days of the start of treatment and must agree to use an effective method of contraception during the trial

Exclusion Criteria:

* Untreated concurrent malignancies or malignancies that have been in complete remission for less than one year
* Treatment with strong inhibitors of CYP3A4 for which there are no therapeutic substitutions
* Inflammatory disorders of the gastrointestinal tract, or subjects with GI malabsorption
* HIV positive; known active hepatitis B or C
* Known hypersensitivity to any of the components of PRT811

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
To describe dose limiting toxicities (DLT) of PRT811 | Baseline through Day 21
  Dose limiting toxicities will be evaluated through the first cycle
To determine the maximally tolerated dose (MTD) | Baseline through approximately 2 years
  The MTD will be established for further investigation in participants with solid tumors and gliomas
To determine the recommended phase 2 dose (RP2D) and schedule of PRT811 | Baseline through approximately 2 years
  The RP2D will be established for further investigation in participants with solid tumors and gliomas

SECONDARY OUTCOMES:
To describe the adverse event profile and tolerability of PRT811 | Baseline through approximately 2 years
  Adverse events as characterized by type, frequency, severity, timing, seriousness and relationship to study therapy
To describe the pharmacokinetic profile of PRT811 | Cycle 1 (each cycle is 21 days) on Days 1, 8 and 14. For subsequent cycles, Day 1 of each cycle through the end of study treatment, an average of 6 months
  PRT811 pharmacokinetics will be calculated including the maximum observed plasma concentration
To describe any anti-tumor activity of PRT811 | Baseline through approximately 2 years
  Anti-tumor activity of PRT811 will be based on the measurement of objective responses

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Yale- New Haven Hospital- Yale Cancer Center, New Haven, Connecticut
  - Christiana Care Health Services, Christiana Hospital, Newark, Delaware
  - Florida Cancer Specialists, Lake Mary, Florida
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - The Ohio State University and Wexner Medical Center, Columbus, Ohio
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee

REFERENCES:
- [Derived] Barry A, Samuel SF, Hosni I, Moursi A, Feugere L, Sennett CJ, Deepak S, Achawal S, Rajaraman C, Iles A, Wollenberg Valero KC, Scott IS, Green V, Stead LF, Greenman J, Wade MA, Beltran-Alvarez P. Investigating the effects of arginine methylation inhibitors on microdissected brain tumour biopsies maintained in a miniaturised perfusion system. Lab Chip. 2023 May 30;23(11):2664-2682. doi: 10.1039/d3lc00204g. PMID 37191188